CLINICAL TRIAL: NCT05650567
Title: A Phase IIa, Randomized, Parallel, Double-Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Enpatoran in Dermatomyositis and Polymyositis Participants Receiving Standard of Care (NEPTUNIA)
Brief Title: Study of M5049 in DM and PM Participants (NEPTUNIA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on interim analyses for futility
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS200569_0041; 2022-501351-82-00 (Other: EUCT number)
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Dermatomyositis; Polymyositis
Keywords: Toll-like Receptor 7; Toll-like Receptor 8; Anti-synthetase syndrome; Idiopathic immune myopathies; Myositis; M5049
MeSH Terms: conditions — Dermatomyositis; Polymyositis; Myositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-blind Placebo Controlled (DBPC) Period: M5049 high dose (Experimental)
  Interventions: Drug: M5049 high dose
- DBPC Period: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Open Label Extension (OLE) Period: M5049 high dose (Experimental)
  Interventions: Drug: M5049 high dose

INTERVENTIONS:
Drug: M5049 high dose — Participants will receive film-coated tablets of M5049 at a high dose orally, twice daily up to 24 weeks.
  Other Names: Enpatoran
  Arms: Double-blind Placebo Controlled (DBPC) Period: M5049 high dose; Open Label Extension (OLE) Period: M5049 high dose
Drug: Placebo — Participants will receive placebo matched to M5049 orally, twice daily up to 24 weeks.
  Arms: DBPC Period: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of orally administered M5049 in idiopathic inflammatory myopathies, specifically dermatomyositis (DM) and polymyositis (PM) participants for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable or definite DM or PM as per 2017 ACR/EULAR classification criteria, with positive autoantibody status. Anti-synthetase syndrome (ASyS) participants that meet classification criteria are allowed
* Active disease on standard of care (SoC), must meet 1 of the criteria within 6 months prior to Screening: Pathological evidence of active myositis in muscle biopsy; Evidence of active myositis by Electromyography (EMG); Magnetic resonance imaging (MRI) with evidence of active myositis; or any muscle enzyme greater than or equal to (>=) 4 × upper limit of normal (ULN) at time of Screening; Active PM/DM skin rash as per cutaneous dermatomyositis area and severity index-A (CDASI-A) >= 7 at time of Screening
* Minimum disease severity defined by: moderate to severe myopathy with manual muscle testing-8 (MMT-8) >= 80 and less than or equal to (<=) 142 AND at least 2 of the following core set measures (CSM) abnormalities: Patient Global Activity (PtGA) >= 2 centimeters (cm); Physician Global Activity (PGA) derived from myositis disease activity assessment tool (MDAAT) >= 2 cm; Extramuscular Activity Assessment derived from MDAAT >2 cm; At least 1 muscle enzyme > 1.5 times ULN; health assessment questionnaire-disability index (HAQ-DI) >= 0.25
* Stable doses of oral corticosteroids (CS) and/or maximum of 1 non-corticosteroid immunosuppressive/immunomodulatory medications (methotrexate, 6 mercaptopurine, sulfasalazine, mycophenolate mofetil or sodium, azathioprine, leflunomide, cyclosporine, oral tacrolimus) for DM or PM
* Participants have a body mass index (BMI) lower or Equal to 40.0 kilograms per square meter (kg/m^2)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Primary diagnosis of inclusion body myositis (IBM), malignancy-associated myositis (defined as diagnosis of myositis within 3 years of cancer), immune mediated necrotizing myopathy (IMNM) with a biopsy characterized as necrotizing biopsy or IMNM with positive anti-signal recognition particle antibody (SRP) or anti 3-hydroxy-3-methylglutaryl-coenzyme A reductase (HMGCR) auto antibodies. Participants with anti-transcription intermediary factor 1 (TIF1) gamma antibody or newly diagnosed (within 1 year) anti MDAT5 antibody should have had adequate screening for cancer within 12 months of Day 1. Adequate screening of cancer is defined as up-to-date age and gender appropriate screening as per national guidelines
* Primary diagnosis of juvenile DM, or adult participants previously diagnosed with juvenile DM
* Any other active concurrent connective tissue disease associated with inflammatory myopathy in the Investigator's opinion. Eligibility of participants with diagnosis of concurrent connective tissue disease(s) will be reviewed and approved by an idiopathic inflammatory myopathies (IIM) expert committee
* Severe interstitial lung disease defined as supplemental oxygen required at rest, or forced vital capacity (FVC) of <60 percent (%) predicted. Participants within 1 year of PM/DM diagnosis and anti-MDA5 antibody, should have been evaluated for interstitial lung disease (ILD) with high resolution computed tomography (HRCT) Chest
* Any uncontrolled disease (for example [e.g.], severe respiratory, cardiovascular, gastrointestinal, neurological, psychiatric, hematological, metabolic [including thyroiditis with increased/decreased thyroid stimulating hormone (TSH)], renal [Estimated glomerular filtration rate < 40 milliliter per minute/1.73 m^2 as calculated by the Modification of Diet in Renal Disease equation by the central laboratory], hepatic, endocrine/reproductive organ disease) other than DM/PM, that in the Investigator's or Sponsor/designee's opinion constitutes an inappropriate risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
DBPC Period: American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Total Improvement Score (TIS) at Week 24 | at Week 24
DBPC Period: Number of Participants with Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and Adverse Events of Special Interest (AESIs) | up to Week 26
DBPC Period: Number of Participants with Clinically Significant Changes from Baseline in Laboratory Parameters, Vital Signs and 12-Lead Electrocardiogram (ECG) Measurements | up to Week 26

SECONDARY OUTCOMES:
DBPC Period: Number of Participants with American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Total Improvement Score (TIS) Greater Than or Equal to (>=) 20, >= 40 and >= 60 | Week 16 and Week 24
DBPC Period: Total Improvement Score (TIS) | Week 4 up to Week 20
DBPC Period: Mean Score for Core Set Measures (CSM) from Week 4 up to Week 24. | Week 4 up to Week 24
DBPC Period: Percent Change from Baseline in Most Abnormal Muscle-associated Enzyme at Weeks 4, 8, 12, 16, 20 and 24 | Baseline, Weeks 4, 8, 12, 16, 20 and 24
DBPC Period: Absolute Change from Baseline in the Core Set Measures (CSM) at Weeks 4, 8, 12, 16, 20 and 24' | Baseline, Weeks 4, 8, 12, 16, 20 and 24
DBPC Period: Percent Change from Baseline in Core Set Measures (CSM) at Weeks 4, 8, 12, 16, 20 and 24' | Baseline, Weeks 4, 8, 12, 16, 20 and 24
DBPC Period: Number of Participants with International Myositis Assessment and Clinical Studies (IMACS) Response | Week 16 and Week 24
DBPC Period: Change from Baseline in Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) A and CDASI-D at Weeks 4, 8, 12, 16, 20 and 24 | Baseline, Weeks 4, 8, 12, 16, 20 and 24
DBPC Period: Percent Change from Baseline in Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) A and CDASI-D at Weeks 4, 8, 12, 16, 20 and 24 | Baseline, Weeks 4, 8, 12, 16, 20 and 24
DBPC Period: Change from Baseline in Investigator's Global Assessment (IGA) Skin Activity Score at Weeks 4, 8, 12, 16, 20 and 24 | Baseline, Weeks 4, 8, 12, 16, 20 and 24
DBPC Period: Percent Change from Baseline in Investigator's Global Assessment (IGA) Skin Activity Score at Weeks 4, 8, 12, 16, 20 and 24 | Baseline, Weeks 4, 8, 12, 16, 20 and 24
OLE Period: Number of Participants with Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and Adverse Events of Special Interest (AESIs) | up to Week 50
OLE Period: Number of Participants with Clinically Significant Changes from Baseline in Laboratory Parameters, Vital Signs and 12-Lead Electrocardiogram (ECG) Measurements | up to Week 50

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (31):
- United States (13):
  - Neuromuscular Research Center, Phoenix, Arizona
  - HonorHealth Research Institute - Bob Bove Neuroscience Institute-Neuroscience Research, Scottsdale, Arizona
  - Mayo Clinic Scottsdale (6365), Scottsdale, Arizona
  - Barbara Davis Center, Aurora, Colorado
  - HMD Research LLC, Orlando, Florida
  - Bolanos Clinical Research, Pembroke Pines, Florida
  - Augusta University-Rheumatology, Augusta, Georgia
  - Johns Hopkins University - Department of Medicine, Division of Rheumatology, Baltimore, Maryland
  - University of Minnesota-Dermatology, Minneapolis, Minnesota
  - University of Kansas Medical Center-Neuromuscular, Kansas City, Missouri
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Austin Neuromuscular Center, Austin, Texas
  - Nerve and Muscle Center of Texas-Clinical research, Houston, Texas
- Institute of Rheumatology - Rheumatology, Prague, Czechia
- Greece (3):
  - Hippokration Hospital - 2nd Department of Medicine and Laboratory, Athens
  - National and Kapodistrian University of Athens (Egnitio Hospital), Athens
  - University General Hospital of Larissa, Larissa
- Italy (5):
  - Azienda Ospedaliero Universitaria Policlinico G. Rodolico-San Marco Di Catania (Vittorio Emanuele) - Reumatologia, Catania
  - Azienda Ospedaliero-Universitaria Policlinico G. Rodolico-San Marco Di Catania, Catania
  - Azienda Usl Toscana Centro, Florence
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Fondazione Policlinico Universitario A. Gemelli-IRCCS, UCSC - Scienze Mediche e Chirurgiche, Rome
- Instytut Reumatologii im. Eleonory Reicher - Department of Connective Tissue Diseases, Warsaw, Poland
- Spain (3):
  - CHUAC - Complexo Hospitalario Universitario A Coruña - Rheumatology, A Coruña
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid - Rheumatology Department, Madrid
- United Kingdom (5):
  - Doncaster Royal Infirmary (3466), Doncaster
  - Royal Free London NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust- Neuromuscular Diseases, London
  - Salford Royal Hospital, Barnes Clinical Research Facility, Salford
  - Royal Wolverhampton Hospitals (6493), Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: https://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200569_0041
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html